CLINICAL TRIAL: NCT04781270
Title: mFOLFOXIRI Plus Bevacizumab Versus mFOLFOX6 Plus Bevacizumab for the First Line Treatment of RAS Mutant Unresectable Colorectal Liver-limited Metastases
Brief Title: mFOLFOXIRI+Bev vs. mFOLFOX6+Bev for RAS Mutant Unresectable Colorectal Liver-limited Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BECOME2
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Carcinoma; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mFOLFOXIRI+Bev (Experimental): Patients will receive mFOLFOXIRI plus bevacizumab once every two weeks as the first-line treatment.
  Drug: mFOLFOXIRI plus Bevacizumab Bevacizumab (5 mg/kg on day 1) plus mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 165 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1). A local MDT will assess the efficiency every 4 cycles of the treatment. The maximum period of conversion therapy is 12 cycles.
  Interventions: Drug: mFOLFOXIRI regimen; Drug: Bevacizumab
- mFOLFOX6+Bev (Active Comparator): Patients will receive mFOLFOX6 plus bevacizumab once every two weeks as the first-line treatment.
  Drug: mFOLFOX6 Plus Bevacizumab mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1). A local MDT will assess the efficiency every 4 cycles of the treatment. The maximum period of conversion therapy is 12 cycles.
  Interventions: Drug: mFOLFOX regimen; Drug: Bevacizumab

INTERVENTIONS:
Drug: mFOLFOXIRI regimen — oxaliplatin 85 mg/m2, irinotecan 165 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1
  Arms: mFOLFOXIRI+Bev
Drug: mFOLFOX regimen — oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1
  Arms: mFOLFOX6+Bev
Drug: Bevacizumab — 5 mg/kg on day 1

SUMMARY:
Colorectal cancer patients with initially unresectable liver-only metastases may be cured after downsizing of metastases by conversion therapy. However, the optimal regimen of conversion therapy for RAS mutant patients has not been defined.

In this study colorectal cancer patients with initially unresectable liver-only metastases, as prospectively confirmed by a local multidisciplinary team (MDT) according to predefined criteria, will be tested for RAS and BRAF tumor mutation status. Patients with RAS mutant and BRAF wild type will be randomised between modified FOLFOXIRI (mFOLFOXIRI) plus bevacizumab and modified FOLFOX6 (mFOLFOX6) plus bevacizumab. Patient imaging will be reviewed for resectability by MDT, consisting of at least one radiologist and three liver surgeons every assessment. MDT review will be performed prior to randomization as well as during treatment, as described in the protocol.

DETAILED DESCRIPTION:
Patients will be stratified for primary tumor location (right-sided or left sided), numbers of liver metastases (<5 or ≥5) and primary tumor resected or unresected.

Patients with RAS mutated primary tumors will be randomized between mFOLFOXIRI plus bevacizumab (Bevacizumab 5 mg/kg in 15-30 minutes i.v., followed by irinotecan 165 mg/m^2 i.v. in 60 minutes, followed by oxaliplatin 85 mg/m^2 i.v. together with leucovorin 400 mg/m^2 i.v. in 120 minutes, followed by continuous infusion of 5-fluorouracil 2400 mg/m^2 in 46 hours, every 2 weeks) or mFOLFOX6 plus bevacizumab (Bevacizumab 5 mg/kg in 15-30 minutes i.v., followed by oxaliplatin 85 mg/m^2 i.v. together with leucovorin 400 mg/m^2 i.v. in 120 minutes, followed by bolus 5FU 400 mg/m^2, all on day 1, followed by continuous infusion of 5-fluorouracil 2400 mg/m^2 in 46 hours, every 2 weeks).

Patients will be evaluated every 8 weeks by MRI or CT scan for disease status. The assigned systemic treatment should be continued for at least 6 months or earlier in case of resectability, progression of disease, unacceptable toxicity, or patient refusal. If after 6 months MDT concludes that the patient is still not resectable, it is highly unlikely that resectability will be achieved at all. Therefore the chemotherapy regimen may be reconsidered after 6 months of treatment. These patients will continue with bevacizumab plus fluoropyrimidine until progression or unacceptable toxicity.

In patients who will become resectable and undergo secondary surgery of liver metastases, the total duration of preoperative and postoperative treatment together should be 6 months. However, in these patients mFOLFOXIRI should not be continued after surgery and replaced by mFOLFOX6. Bevacizumab will continued after surgery for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal adenocarcinoma;
* Age ≥ 18 years and ≤75 years;
* Simultaneous liver-limited metastases;
* Initially unresectable liver metastases determined by a local MDT;
* RAS mutation and BRAF V600E wild-type;
* At least one measurable liver metastasis;
* Initially resectable primary tumor or primary tumor already resected;
* World Health Organization (WHO) performance status 0-1;
* Life expectancy ≥ 3 months;
* Adequate hematologic function: absolute neutrophil count (ANC)≥1.5×109/l, platelets≥100×109/l, and hemoglobin(HB) ≥ 9g/dl;
* Adequate liver and renal function: total bilirubin ≤2.0 mg/dl, serum transaminases ≤ 5x upper limit of normal(ULN), and serum creatinine ≤ 1.5x ULN and creatinine clearance ≥ 30 ml/min;
* Written informed consent.

Exclusion Criteria:

* Previous systemic treatment for metastatic disease;
* Previous surgery for metastatic disease;
* Extrahepatic metastases;
* Unresectable primary tumor;
* Major cardiovascular events (myocardial infarction, severe/unstable angina, congestive heart failure, CVA) within 12 months before randomisation;
* Acute or subacute intestinal obstruction;
* Second primary malignancy within the past 5 years;
* Drug or alcohol abuse;
* No legal capacity or limited legal capacity;
* Pregnant or lactating women;
* Uncontrolled hypertension, or unsatisfactory blood pressure control with ≥3 antihypertensive drugs;
* Peripheral neuropathy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
conversion resection rate | up to 6 months
  R0 resection rate upon conversion treatment with chemotherapy plus bevacizumab

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  from the first day of assigned treatment to death or last known to be alive
Progression-free survival (PFS) | up to 2 years
  from the first day of assigned treatment to progression or death whichever comes first
Toxicity (AE) | up to 6 months
  Patients will be evaluated for Adverse Events at the start of each treatment cycle according to CTCAE version 5.0
postoperative complication | After surgery during one month
  Patients will be evaluated for surgical morbidity during 1 month. Postoperative morbidity will be scored according 'Clavien-Dindo Grade'.
overall response | up to 6 months
  Response according to RECIST 1.1
proportion of no evidence of disease | up to 6 months
  Response according to RECIST 1.1
Best deepness of response | up to 6 months
  The maximum tumor shrinkage rates by Response Evaluation Criteria in Solid Tumors (RECIST) throughout the treatments
Early tumor shrinkage | at 8 weeks
  The rates of tumor shrinkage by RECIST at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China